CLINICAL TRIAL: NCT00300911
Title: A Study of PPAR-Gamma Agonist-Rosiglitazone for Determining Cardiac Adverse Effects in Type 2 Diabetic Patients
Brief Title: Effects of Rosiglitazone on Plasma BNP Levels and Left Ventricular Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA04/164
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2006-03-10 (Estimated); Status verified 2005-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Natriuretic Peptide, Brain; Heart Failure, Congestive
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure

INTERVENTIONS:
Drug: Rosiglitazone(drug), cardiac adverse effects

SUMMARY:
The present study aimed to evaluate the effect of rosiglitazone treatment on cardiac function compared with metformin

DETAILED DESCRIPTION:
Large scale clinical trials have reported fluid retention and increase in plasma volume (6% to 7%) with glitazone therapy, with an increased incidence of peripheral edema occuring in 2% to 5% patients. Some evidence suggests that this effect may be related to increased endothelial cell permeability induced by glitazones therapy. Others report that glitazones may interfere with renal hemodynamics. In controlled clinical trials, the frequency of new onset congestive heart failure was very low in glitazones treated patients. The incidence of congestive heart failure is higher in patients receiving combination therapy with insulin and glitazones. Only few studies compared rosiglitazone and metformin on cardiac safety. Recently a study reported a reversible increase in endothelial cell permeability to albumin in cultured pulmonary arterial cells treated with rosiglitazone. To our knowledge, there is not any clinical study published for showing the reversibility of the cardiac adverse effects if the rosiglitazone treatment is continued.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treated with oral hypoglycemic agents or diet only
* Without any symptom or finding of heart failure
* Normal liver enzymes and renal functions

Exclusion Criteria:

* Any known coronary artery disease, congestive hearth failure, renal disease or liver disease
* Any treatment for heart failure or diuretics for any reasons.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-12

PRIMARY OUTCOMES:
Plasma Brain Natriuretic Peptide levels, echocardiographic measurements were made before the treatment and repeated after three months and six months of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin T Kemal, MD, Study Director — Medical Doctor, Internal Medicine
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Niemeyer NV, Janney LM. Thiazolidinedione-induced edema. Pharmacotherapy. 2002 Jul;22(7):924-9. doi: 10.1592/phco.22.11.924.33626. PMID 12126225
- [Background] Wooltorton E. Rosiglitazone (Avandia) and pioglitazone (Actos) and heart failure. CMAJ. 2002 Jan 22;166(2):219. No abstract available. PMID 11826947
- [Background] Idris I, Gray S, Donnelly R. Rosiglitazone and pulmonary oedema: an acute dose-dependent effect on human endothelial cell permeability. Diabetologia. 2003 Feb;46(2):288-90. doi: 10.1007/s00125-002-1008-1. Epub 2003 Feb 12. PMID 12627329
- [Background] Maeda K, Tsutamoto T, Wada A, Hisanaga T, Kinoshita M. Plasma brain natriuretic peptide as a biochemical marker of high left ventricular end-diastolic pressure in patients with symptomatic left ventricular dysfunction. Am Heart J. 1998 May;135(5 Pt 1):825-32. doi: 10.1016/s0002-8703(98)70041-9. PMID 9588412
- [Background] Lubien E, DeMaria A, Krishnaswamy P, Clopton P, Koon J, Kazanegra R, Gardetto N, Wanner E, Maisel AS. Utility of B-natriuretic peptide in detecting diastolic dysfunction: comparison with Doppler velocity recordings. Circulation. 2002 Feb 5;105(5):595-601. doi: 10.1161/hc0502.103010. PMID 11827925
- [Background] Ogawa S, Takeuchi K, Ito S. Plasma BNP levels in the treatment of type 2 diabetes with pioglitazone. J Clin Endocrinol Metab. 2003 Aug;88(8):3993-6. doi: 10.1210/jc.2002-021765. PMID 12915698